CLINICAL TRIAL: NCT04047394
Title: An Open Label, Single-dose, Dose-increasing Study to Assess the Safety, Tolerability, PK and Preliminary PD of PEGylated Recombinant Candida Urate Oxidase (SSS11) for Injection in Chinese Healthy Adult Volunteers
Brief Title: A Study to Determine the Safety, Tolerability, PK and Preliminary PD of SSS11 in Chinese Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-SSS11-UND-Ⅰ-02
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEGylated recombinant candida urate oxidase (Experimental): Participants will be administered with 2mg, 3mg, 4.5mg, 6mg, 8mg, 10mg once by Intravenous injection. Subjects will be followed for 56 days.
  Interventions: Drug: PEGylated recombinant candida urate oxidase

INTERVENTIONS:
Drug: PEGylated recombinant candida urate oxidase — PEGylated recombinant candida urate oxidase is a combination of 20kDa linear polyethylene glycol (PEG) linked to Candida utilis recombinant uricase by succinimide succinate
  Other Names: SSS11

SUMMARY:
To evaluate the safety, tolerability, PK and preliminary PD of SSS11 for injection in chinese healthy adult volunteers.

DETAILED DESCRIPTION:
This is a phase I, open label, single-dose, dose-increasing study to assess the safety, tolerability and PK characteristics of healthy humans after injection of SSS11, provide a reference for subsequent clinical studies and give preliminary assessment of the immunogenicity and PD of SSS11.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age range between 18 and 45 years old (inclusive), male or female
* In good health (no significant clinical symptoms or abnormal laboratory test results without clinical significance)
* BMI within the range between 19 and 28 kg/m2 (inclusive)
* Voluntarily sign the written informed consent
* Be able to understand and comply with the requirements of clinical protocols, expected to complete the whole trial process
* Subjects achieving full recovery if had the surgical treatment

Exclusion Criteria:

* Subjects cannot tolerate intravenous injection
* Allergies or previous history of drug allergy, or allergic history of PEG-drugs, or previous history of allergies to two or more substances
* Any abnormalities detected in three allergen tests (Special allergen screening - mixed mould, total IgE assay, special allergen screening - HX2)
* Subjects having anti- PEG antibody
* Taking any medicine before enrollment, and the regimen was less than five half-life periods or 4 weeks (Subject to the longest of the two)
* Has a history of vaccination within 12 weeks before enrollment, or intend to receive vaccines during the study
* Taking any other clinical trials within 12 weeks before enrollment,or have used similar drugs to the study drug
* Having a history of blood donation within 12 weeks before enrollment
* Having a history of glucose-6-phosphate dehydrogenase (G6PD) deficiency or abnormal G6PD detection
* Having a history of catalase deficiency or evidence that individuals meet the criteria for catalase deficiency
* Having a history of serious diseases, including but not limited to digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, immune system diseases and metabolic abnormalities
* Having abnormalities and clinical significances in laboratory tests (blood routine, urine routine, blood biochemistry, etc.) and electrocardiogram findings within two weeks before enrollment
* The HBsAg, anti-HIV, anti-HCV and treponema pallidum antibody were positive
* The female within lactation, pregnancy, or having birth plan within 24 weeks
* Blood pregnancy test was positive(female)
* Male subjects who did not take effective contraception or their spouse plan to be born within 24 weeks
* Disabled person in mental or law
* Subjects having a history of alcohol abuse within 24 weeks prior to screening, equal to exceed 14 unit alcohol per week (1 unit = 12 ounces or 360 mL of beer, 1.5 ounces or 45 mL of 40% alcohol, 5 ounces or 150 mL of wine)
* Smoking more than 5 cigarettes per day within 24 weeks before screening
* Those who have had halo and fainting history
* Drug abuse test or alcohol test was positive
* Drinking more than 1L of tea, coffee and/or caffeinated beverages daily
* Those who do not understand the content of informed consent and other those who do not meet the criteria for trial inclusion
* Participants who researchers believe are not suitable (such as infirmity, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From the day signing in informed consent form to the day 56 post-dose
  Number of subjects with Adverse events (AEs)
DLT | From day 1 to day 56
  Dose-LimitingToxicity of SSS11
Cmax | From beginning of drug administration to day 56
  Maximum plasma concentration (Cmax) of single dose SSS11
Tmax | From beginning of drug administration to day 56
  Peak plasma time [tmax] of single dose SSS11
AUC | From beginning of drug administration to day 56
  Area under the plasma concentration versus time curve (AUC) of single dose SSS11

SECONDARY OUTCOMES:
Anti-urate oxidase antibody | From pre-dose on week 2 up to week 1, 2, 4 and 7 post-dose.
  The immunogenicity of SSS11 was assessed in subjects by detecting the anti-urate oxidase antibody.
Uric acid levels in blood | From beginning of drug administration to day 56
  This parameter was used to evaluate the PD of SSS11 in healthy humans.
Uric acid levels in urine | From beginning of drug administration to day 6
  This parameter was used to evaluate the PD of SSS11 in healthy humans.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided